CLINICAL TRIAL: NCT03224143
Title: Doll Therapy Efficacy for People With Dementia Living in Nursing Homes: a Randomized Single-blind Controlled Trial
Acronym: ADTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Collaborators: Fondazione Golgi Cenci (Other); University of Turin, Italy (Other); Gruppo Doll Therapy Ticino (Unknown); Case per Anziani Canton Ticino (Unknown); Centro di Terapia Cognitiva, Como (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE3140 BASEC2016-01992
Record Dates: First submitted 2017-03-15; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Dementia
Keywords: dementia; doll therapy; attachment
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Each participant will undergo daily sessions of DTI or SI, lasting an hour at most, led by a trained professional caregiver. The DTI involves the presentation of a doll produced by a Swedish brand conceived for Doll Therapy use. The SI group will attend similar daily sessions, but in place of the doll, it will be presented with a non-anthropomorphic object, i.e., a soft foam rubber cube covered with a coloured and velvety textile. The 1st and 30th session of all participants will be videotaped by a trained psychologist as described below. The experimental protocol is described in detail in Pezzati et al. (2014) and it is structured with the goal of recreating a situation of (1) separation from a known figure and (2) interaction with the environment in order to partially recreate the prototypical phases of the "Strange situation" (Ainsworth et al., 1978).
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, the psychologist who will administer the NPI-NH will not be aware of the arm to which the subjects belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doll Therapy Intervention (DTI) (Experimental): The DTI involves the presentation of a doll produced by a Swedish brand and conceived for Doll Therapy use. It is designed to recreate the sensation of touching, looking and holding a child in the arms. The doll presentation involves five standard steps:
  1. A nurse (whom the patient knows) accompanies the patient in the room and invites her to sit on the chair.
  2. The nurse presents the object (doll or cube) to the patient.
  3. The nurse leaves the patient alone with the object.
  4. Interaction with the object: it lasts 3 minutes starting from the moment when the nurse leaves the room. This phase is interrupted if the patient drops the object before the time limit.
  5. The nurse returns into the room and takes back the object.
  Interventions: Behavioral: Doll Therapy Intervention
- Active control group (SI) (Active Comparator): The SI involves the presentation of a non-anthropomorphic object, a soft foam rubber cube covered with a coloured and velvety textile. The procedure is the following:
  1. A nurse (whom the patient knows) accompanies the patient in the room and invites her to sit on the chair.
  2. The nurse presents the cube to the patient.
  3. The nurse leaves the patient alone with the cube.
  4. Interaction with the cube: it lasts 3 minutes starting from the moment when the nurse leaves the room. This phase is interrupted if the patient drops the object before the time limit.
  5. The nurse returns into the room and takes back the cube.
  Interventions: Behavioral: active control group (SI)

INTERVENTIONS:
Behavioral: Doll Therapy Intervention — Daily sessions, lasting an hour, will take place in a room known to patients (P). The only people in the room will be a nurse (N) and the researcher with video-tape, never interacting with P. The procedure is: the N will accompany the P in the room and the P will take a seat. The N will put the doll in front of the P and will say "Good morning Mr./Mrs....look", with a quiet voice. If the P will not take it at the first attempt, the N will sit down in front of her holding the doll in the arms and will wait for 2 minutes. The N will invite the PWD again. If the P will not take the doll after the second request, the N will not insist and she will leave. If the doll will be taken, the N will leave the P and say "I have to go, goodbye Mr./Mrs. . . ..". The gaze will always be upon the P.
  Arms: Doll Therapy Intervention (DTI)
Behavioral: active control group (SI) — Daily sessions, lasting an hour, will take place in a room known to patients (P). The only people in the room will be a nurse (N) and the researcher with video-tape, never interacting with P. The procedure is: the N will accompany the P in the room and the P will take a seat. The N will put the cube in front of the P and will say "Good morning Mr./Mrs....look", with a quiet voice. If the P will not take it at the first attempt, the N will sit down in front of her holding the cube in the arms and will wait for 2 minutes. The N will invite the PWD again. If the P will not take the cube after the second request, the N will not insist and she will leave. If the cube will be taken, the N will leave the P and say "I have to go, goodbye Mr./Mrs. . . ..". The gaze will always be upon the P.
  Arms: Active control group (SI)

SUMMARY:
This study is a randomized single-blind controlled trial with parallel arms.The present study is based on that previously published by Pezzati and collegues (2014) and it is part of a larger project focusing on Doll Therapy dissemination in Canton Ticino through team training and supervision and guidelines definition that led to the establishment of the Ticino Doll Therapy Group with support of the Canton Office for elderly and home care.

The first hypothesis regards the 30 days-effectiveness efficacy of the Doll Therapy intervention in reducing symptoms of behavioral disorders (BPSD) that appear in stressful situations (as in the case of a separation from a professional caregiver) and in reducing stress as perceived by the treating physician. Another issue to be investigated is whether the typical way in which a person manifested attachment behaviors during own life (classified in three types of mental states: secure, insecure and unresolved) is associated, once this person is in an advanced stage of dementia, with caregiving behaviors of the PWD during the doll presentation (i.e. caressing the object, talking to it and smiling).

DETAILED DESCRIPTION:
Primary goals The primary goal of the present study is to evaluate the efficacy of Doll Therapy Intervention (DTI) versus a Sham Intervention (SI), on behavioral and psychiatric symptoms of PWD living in a nursing home. Outomes will be measured with the Italian version of Neuropsychiatric Inventory-Nursing Home. It is expected an improvement in terms of a decrease in NPI-NH total score.

We will also assess the efficacy of DTI versus SI, on professional caregivers distress ratings related to behavioral and psychiatric symptoms of PWD. It will be measured with the Italian version of NPI-NH. It is expected an improvement in terms of a decrease in NPI-NH distress total score.

It will also assess the efficacy of DTI versus SI, on cognitive and physiological status of PWD. The first will be recorded as the presence or absence of exploratory and caregiving behaviors on an observational grid expressly conceived for this purpose (Grid 2, Appendix). It is expected an improvement in terms of an increase of the number and duration of exploratory and caregiving behaviors. The efficacy of DTI versus SI on physiological status of PWD will be measured by assessing blood pressure (systolic and diastolic), heart rate, and salivary cortisol that are biomarkers of acute stress. It is expected an improvement in terms of a decrease in these parameters.

All evaluations will be performed at baseline (T0) and thirty days later (T1). Secondary goal The secondary goal is to evaluate the stability of attachment behaviors of the PWD through the adminstration of the Adult Attachment Interview to the patients' offspring after conclusion of interventions. It is expected to find an association between the attachment style of the PWD and caregiving behaviors during the doll presentation (i.e. caressing the object, talking to it and smiling). Such behaviors are recorded in an observational grid expressely conceived for this purpose.

These observations will allow the investigators to test wether a relationship between present and past attachment style of PWD and between attachment styles and participant response to doll therapy exist. Investigators expect that PWD with a previous secure attachment style will accept the doll and will show caregiving behaviors, while the PWD with insecure attachment style will show, especially during the first contacts, rejection, avoidance of the doll or excessive caregiving reactions towords the doll. Investigators also expect that PWD with unresolved attachment style will show inconsistent responses to the presentation of the doll, with approaching and rejecting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* • presence of moderate to severe dementia, assessed with Global Deterioration Scale (GDS 4-7);

  * presence of at least one behavioral and psychiatric symptom (BPSD) in addition to depression or apathy (Lai, 2014) assessed with the NPI-NH;
  * female gender;
  * admission in the nursing home at least 3 months before;
  * no previous Doll Therapy exposure;
  * presence of a daughter or a son, as a family caregiver

Exclusion Criteria:

* male gender
* presence of previous comorbid mental disorders, such as major depression, bipolar disorders and schizophrenia;
* inability to sit comfortably on a chair or limitations in mobility of the arms;
* presence of acute clinical conditions interfering with the participation to the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-02-16 (Estimated); Study Completion 2020-02-16 (Estimated)

PRIMARY OUTCOMES:
Behavioral and psychiatric symptoms | from baseline (T0) to 30 days since the beginning of intervention (T1)
  A decrease of the behavioral and psychiatric symptoms of patient measured as the net change in the total scores of the Nursing Home version of NPI (NPI-NH total score) from baseline to post-intervention. It is expected a significant difference in NPI-NH total scores between experimental and active control group. The NPI-NH will be administered to the team of the nursing home by a trained blinded psychologist. The NPI-NH is specifically designed for interviewing professional care facility staff.
Professional caregiver distress | from baseline (T0) to 30 days since the beginning of intervention (T1).
  A decrease of the professional caregiver distress ratings related to behavioral and psychiatric symptoms of patient. It is measured as the net change in the distress total score of the Nursing Home version of NPI (NPI-NH-D total score) from baseline to post-intervention.
Interaction with the object | from baseline (T0) to 30 days since the beginning of intervention (T1)
  An increase of the duration (expressed in seconds) of the interaction with the object: it is expected a significant difference in duration between experimental and control group. This measure is recorded by professional caregivers during the daily sessions of DTI or SI.
Salivary cortisol | from the time immediately before to 15 minutes after each daily sessions of DTI or SI
  Salivary cortisol is a biomarker of stress, and its secretion is the final product of the activation of stress-response mechanisms, specifically the hypothalamic-pituitary-adrenal axis. It is expected a significantly different decrease of the concentration of salivary cortisol between experimental and control group.
Blood pressure | ffrom the time immediately before to 15 minutes after each daily sessions of DTI or SI
  A significantly different decrease of the blood pressure (systolic and diastolic) of the patients between experimental and control group.
Heart rate | from baseline (T0) to 30 days since the beginning of intervention (T1).
  A significantly different decrease of the heart rate of the patients between experimental and control group.

SECONDARY OUTCOMES:
association between the pre-morbid attachment style of PWD and the response to DTI | after 30 days since the beginning of intervention (T1)
  The Adult Attachment Interview (AAI) is a semi-structured interview administered to children of the patients in the DTI group in order to identify mental states related to attachment style. Since a correspondence of 75% between the individual's attachment and that of the own children has been reported, the AAI is a useful instrument to recognize the pre-morbid attachment style of patient. It is video-recorded, and the labeling of the answers is carried out by an external trained and authorized psychologist. it is expected a significant association between the pre-morbid attachment style of patient and the response to DTI.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pezzati, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland
Locations (1):
- SUPSI, Manno, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data transcription and data entry will be under responsibility of SUPSI. Data ownership will remain with SUPSI who signed a contract of availability to the use for the purposes of research, dissemination of results and their publication. All visual and paper material will be stored at SUPSI in closets and filing cabinets fitted with keys. Information recorded on paper will be promptly transferred in a specifically designed password-protected electronic archive or database; access to the personal computer containing the electronic implementation will be protected by an access key. In the database, each subject will be associated to an participant code without identity record, which will be stored separately and protected by password known only to the research manager or her delegate. The code will constitute the key linkage between subjects' identity record and the information obtained during the Doll Therapy study.

REFERENCES:
- [Background] Ainsworth, M., Blehar, M., Waters, E., & Wall, S. (1978). Patterns of attachment. Hills-dale. NJ Eribaum.
- [Background] Bradley JM, Cafferty TP. Attachment among older adults: current issues and directions for future research. Attach Hum Dev. 2001 Sep;3(2):200-21. doi: 10.1080/14616730126485. PMID 11708737
- [Background] Browne CJ, Shlosberg E. Attachment theory, ageing and dementia: a review of the literature. Aging Ment Health. 2006 Mar;10(2):134-42. doi: 10.1080/13607860500312118. PMID 16517488
- [Background] Ellingford, L., Mackenzie, L., & Marsland, L. (2007). Using dolls to alter behavior in people with dementia. Nursing Times, (103), 36-37.
- [Background] George, C., Kaplan, N., & Main, M. (1985). Adult Attachment Interview. (U. of C. Department of Psychology, Ed.)Unpublished manuscript. Berkeley.
- [Background] James IA, Mackenzie L, Mukaetova-Ladinska E. Doll use in care homes for people with dementia. Int J Geriatr Psychiatry. 2006 Nov;21(11):1093-8. doi: 10.1002/gps.1612. PMID 16955418
- [Background] Miesen, B., & Jones, G. (2010). Care-giving in dementia: Contours of a curriculum. Dementia, 9(4), 473-489. http://doi.org/10.1177/1471301210381680
- [Background] Lupien SJ, Lepage M. Stress, memory, and the hippocampus: can't live with it, can't live without it. Behav Brain Res. 2001 Dec 14;127(1-2):137-58. doi: 10.1016/s0166-4328(01)00361-8. PMID 11718889
- [Background] Mitchell G, McCormack B, McCance T. Therapeutic use of dolls for people living with dementia: A critical review of the literature. Dementia (London). 2016 Sep;15(5):976-1001. doi: 10.1177/1471301214548522. Epub 2014 Aug 25. PMID 25160532
- [Background] Pezzati R, Molteni V, Bani M, Settanta C, Di Maggio MG, Villa I, Poletti B, Ardito RB. Can Doll therapy preserve or promote attachment in people with cognitive, behavioral, and emotional problems? A pilot study in institutionalized patients with dementia. Front Psychol. 2014 Apr 21;5:342. doi: 10.3389/fpsyg.2014.00342. eCollection 2014. PMID 24795682
- [Background] van IJzendoorn MH. Adult attachment representations, parental responsiveness, and infant attachment: a meta-analysis on the predictive validity of the Adult Attachment Interview. Psychol Bull. 1995 May;117(3):387-403. doi: 10.1037/0033-2909.117.3.387. PMID 7777645
- [Background] Vreeburg SA, Zitman FG, van Pelt J, Derijk RH, Verhagen JC, van Dyck R, Hoogendijk WJ, Smit JH, Penninx BW. Salivary cortisol levels in persons with and without different anxiety disorders. Psychosom Med. 2010 May;72(4):340-7. doi: 10.1097/PSY.0b013e3181d2f0c8. Epub 2010 Feb 26. PMID 20190128
- [Background] Tamura, T., Nakajima, K., Nambu, M., Nakamura, K., Yonemitsu, S., Itoh, A., … Uno, H. (2001). Baby dolls as therapeutic tools for severe dementia patients. Gerontechnology, 1(2), 111-118.
- [Background] Tsigos C, Chrousos GP. Hypothalamic-pituitary-adrenal axis, neuroendocrine factors and stress. J Psychosom Res. 2002 Oct;53(4):865-71. doi: 10.1016/s0022-3999(02)00429-4. PMID 12377295
- [Background] Quirin M, Gillath O, Pruessner JC, Eggert LD. Adult attachment insecurity and hippocampal cell density. Soc Cogn Affect Neurosci. 2010 Mar;5(1):39-47. doi: 10.1093/scan/nsp042. Epub 2009 Dec 9. PMID 20007241
- [Background] Lai CK. The merits and problems of Neuropsychiatric Inventory as an assessment tool in people with dementia and other neurological disorders. Clin Interv Aging. 2014 Jul 8;9:1051-61. doi: 10.2147/CIA.S63504. eCollection 2014. PMID 25031530
- [Background] Green L, Matos P, Murillo I, Neushotz L, Popeo D, Aloysi A, Samuel J, Craig E, Porter C, Fitzpatrick JJ. Use of dolls as a therapeutic intervention: relationship to previous negative behaviors and pro re nata (prn) Haldol use among geropsychiatric inpatients. Arch Psychiatr Nurs. 2011 Oct;25(5):388-9. doi: 10.1016/j.apnu.2011.05.003. Epub 2011 Jul 12. PMID 21978807
- [Background] Consedine NS, Magai C. Attachment and emotion experience in later life: the view from emotions theory. Attach Hum Dev. 2003 Jun;5(2):165-87. doi: 10.1080/1461673031000108496. PMID 12791565
- [Background] Baranzini F, Grecchi A, Berto E, Costantini C, Ceccon F, Cazzamalli S, Callegari C. [Factor analysis and psychometric properties of the Italian version of the Neuropsychiatric Inventory-Nursing Home in an institutionalized elderly population with psychiatric comorbidity]. Riv Psichiatr. 2013 Jul-Aug;48(4):335-44. doi: 10.1708/1319.14631. Italian. PMID 24056833
- [Derived] Vaccaro R, Ballabio R, Molteni V, Ceppi L, Ferrari B, Cantu M, Zaccaria D, Vandoni C, Ardito RB, Adenzato M, Poletti B, Guaita A, Pezzati R. Doll therapy intervention for women with dementia living in nursing homes: a randomized single-blind controlled trial protocol. Trials. 2020 Feb 3;21(1):133. doi: 10.1186/s13063-020-4050-8. PMID 32014029